CLINICAL TRIAL: NCT07178327
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Administration of LYN101 in Healthy Subjects and Multiple Administrations in Postmenopausal Women With Low Bone Mass
Brief Title: Phase I Clinical Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of LYN101
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai TTM-Bio Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYN101CN001; CTR20253437 (Registry Identifier: National Medical Products Administration)
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteoporotic Fracture
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYN101 (Experimental): In part A, up to 4 single ascending dose cohorts. In part B, one or additional doses for multiple dose cohorts.
  Interventions: Drug: LYN101
- Placebo (Placebo Comparator): Eligible participants will receive the matched placebo via SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LYN101 — In Part A, participants will receive single dose of LYN101 administered as a subcutaneous (SC) injection.
  In Part B, participants will receive multiple doses of LYN101 administered as a SC injection.
  Arms: LYN101
Drug: Placebo — In Part A, participants will receive single dose of the matched placebo administered as a subcutaneous (SC) injection (4 cohorts).
  In Part B, participants will receive multiple doses of the matched placebo administered as a SC injection.
  Arms: Placebo

SUMMARY:
This is a Phase 1, two-part, first-in-human, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single dose of LYN101 in healthy subjects (part A) and multiple doses in postmenopausal women with low bone mass (part B).

DETAILED DESCRIPTION:
The study includes Part A and Part B. Up to four dose levels will be tested in the single ascending dose stage, involving approximately 32 healthy volunteer subjects, with eight subjects per dose level (Part A). After completing Part A, one dose level or additional optional levels will be tested in multiple doses in Part B, enrolling about 12 postmenopausal women with low bone mass. In both Part A and Part B, eligible subjects will be randomized in a 3:1 ratio to receive either LYN101 or a matched placebo.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Part A:

1. Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical study, and sign a written informed consent form.
2. Individuals aged 18 to 65 years (inclusive), regardless of gender;
3. Weight ≥ 50 kg for males or at least 45 kg for females, with a Body Mass Index (BMI) ranging from 18.0 to 30.0 kg/m² (inclusive).
4. Males and females of childbearing potential agree not to plan for childbearing and to use reliable contraceptive measures from the time of signing the written informed consent until 6 months after dosing. They also agree not to donate sperm or ova.

Inclusion Criteria for Part B:

1. Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial, and sign a written informed consent form.
2. Individuals aged 50-70 years (inclusive), female, and ambulatory.
3. Spontaneous amenorrhea lasting for at least two years or bilateral oophorectomy performed at least two years prior. For women under 60 years of age who have undergone hysterectomy but retained their ovaries, or when the status of bilateral oophorectomy is unknown, menopausal status must be confirmed by follicle-stimulating hormone (FSH) levels exceeding 40 mIU/mL or in accordance with the postmenopausal range established by the local laboratory.
4. During the screening process, at least two consecutive vertebrae within the L1-L4 region must be evaluable for DXA BMD assessment, and at least one hip must also be evaluable for DXA BMD assessment.
5. Low bone mass, as measured by Dual Energy X-ray Absorptiometry (DXA) during screening (BMD), shall meet the criteria if any site has a T-score less than -1.0 and greater than -2.5 at the lumbar spine L1-L4, femoral neck, or total hip.

Exclusion Criteria:

Exclusion Criteria for Part A:

1. Systolic blood pressure (SBP) ≥140 mm Hg and/or diastolic blood pressure (DBP) ≥90 mm Hg after at least five minutes of rest during screening assessments.
2. Clinically significant abnormalities observed in the 12-lead ECG at screening include, but are not limited to, a Mean QTcF > 450 ms for males or > 470 ms for females. The measurement is taken while the subject is supine after resting for at least 10 minutes, with three readings obtained at intervals of at least 1 minute. If the mean QTcF exceeds these limits, the ECG measurement should be repeated three times. If the retest results are still abnormal, the subject is excluded.

   PR interval < 120 ms PR interval > 200 ms
3. Clinically significant abnormalities in laboratory tests, chest X-ray, and/or abdominal ultrasound at Screening unless the Investigator determines they are non-interfering.
4. 25-hydroxyvitamin D3 concentration < 20 ng/mL at screening and unwilling to supplement vitamin D.
5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and/or total bilirubin (TBIL) levels exceeding the upper limit of normal (ULN) at screening.
6. International normalized ratio (INR) greater than 1.5 at screening.
7. Corrected serum calcium and phosphorus levels outside the laboratory reference range at Screening (calcium and phosphorus supplements should not be taken for at least 8 hours before measuring serum calcium and phosphorus).
8. Estimated creatinine clearance <60 mL/min (using the Cockcroft-Gault formula) at screening.
9. Any disease that might impact the safety evaluation of the subject or the in vivo process of the investigational product, including the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematopoietic system, metabolic endocrine system, and others.
10. Participation in any other drug or device clinical trials within 30 days or five half-lives (whichever is longer) before screening.
11. Use of prescription drugs within 14 days or five half-lives (whichever is longer) before administering the investigational product, unless the Investigator and Sponsor determine they are non-interfering (e.g., hormonal contraceptives).
12. Use of over-the-counter (OTC) drugs within 7 days or five half-lives (whichever is longer) before administering the investigational product, unless the Investigator and Sponsor determine they are non-interfering.
13. Test results show positive for the hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, Treponema pallidum antibody, or human immunodeficiency virus (HIV) antibody.
14. Use of more than 10 sticks per day of tobacco or nicotine products within the past 30 days before screening.
15. History of alcohol, drug, or substance abuse within the 12 months before screening.
16. Known allergy to human immunoglobulins, the investigational product or its components, calcium preparations, or vitamin D preparations.
17. Receiving a live vaccine (excluding influenza vaccine) within 4 weeks before screening, or planning to receive a live vaccine during the study.
18. Blood donation or blood loss of 400 mL or more within the past thirty days before screening.
19. Pregnant or breastfeeding women.
20. Any condition that, in the investigator's opinion, makes the subject unsuitable for enrollment or may interfere with the subject's participation or completion of the study.

Exclusion Criteria for Part B:

1. Presence of bone metabolic diseases such as hypoparathyroidism, hyperparathyroidism, hypothyroidism, hyperthyroidism, hypopituitarism, hyperprolactinemia, Cushing's syndrome, acromegaly, Paget's disease, rheumatoid arthritis, osteomalacia, among others; individuals with stable hypothyroidism (for at least three months) on thyroid hormone replacement therapy may be eligible for enrollment, provided they meet the following criteria: a TSH level ranging from 4.0 to 10.0 μIU/mL and serum FT4 within the normal range.
2. The following medications that may affect bone metabolism have been received: glucocorticoids (≥ prednisone 5 mg/day or equivalent, taken for at least 10 consecutive days), vitamin K, calcitonin preparations, selective estrogen receptor modulators, sex hormone preparations (excluding vaginal tablets and creams for vaginal use), immunomodulatory agents (such as cyclosporine, tacrolimus, etc.), or methotrexate (excluding calcium and vitamin D supplements) within the past two months; alternatively, bisphosphonates used within the 12 months before screening or used continuously for more than one year within the last two years; or the use of parathyroid hormone (PTH) analogs, anti-RANK ligand (RANKL) antibodies, cathepsin K inhibitors, or anti-Sclerostin antibodies.
3. The individual has a 25-hydroxyvitamin D3 level below 20 ng/mL at screening and has indicated unwillingness to take vitamin D supplements.
4. Estimated creatinine clearance below 60 mL/min (Cockcroft-Gault formula) during screening.
5. Corrected serum calcium levels were outside the laboratory reference range at screening. (Calcium preparations should not be taken for at least 8 hours before measuring serum calcium during screening.)
6. Systolic blood pressure (SBP) is 140 mmHg or higher, and/or diastolic blood pressure (DBP) is 90 mmHg or higher, after at least five minutes of rest during screening.
7. Mean QTcF >470 ms at Screening (measured supine after resting for at least 10 minutes, 3 times with at least 1 minute interval); If the mean QTcF exceeds this limit, repeat the 12-lead ECG measurement 3 times; if the results of the retest are still abnormal, the subject is excluded.
8. Clinically significant cardiovascular, respiratory, digestive, dermatological, urinary, hematological, neurological, psychiatric, or other systemic diseases or laboratory abnormalities, and if the investigator determines the subject is unsuitable for participation.
9. Malignancy within the past 3 years (except completely resected in-situ basal cell or squamous cell skin cancer, cervical carcinoma in situ, or ductal carcinoma in situ of the breast).
10. Known active tuberculosis.
11. Positive for HBsAg, HCV antibody, HIV antibody, or Treponema pallidum antibody. 12. Participation in any other drug or device clinical trials within 30 days or five half-lives (whichever is longer) before screening.

13. Known allergies to human immunoglobulins, the investigational product, its components, calcium supplements, or vitamin D supplements.

14. Receiving a live vaccine (excluding influenza vaccine) within 4 weeks before screening, or planning to receive a live vaccine during the study.

15. History of alcohol, drug, or substance abuse. 16. Fragility fracture within six months before enrollment or when the Investigator considers subjects to be at high risk of fragility fracture requiring treatment with active medications (other than calcium and vitamin D supplements) (Fragility fracture: a fracture occurring under normal or minimal external force due to the inherent fragility of the bone).

17. Any condition that, in the Investigator's opinion, makes the subject unsuitable for enrollment or may interfere with the subject's participation or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-06 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to Day 91 from dosing in part A. Up to 265 from first dosing in part B.
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related during study

SECONDARY OUTCOMES:
Bone turnover markers | Up to Day 91 in part A. Up to 265 in part B.
  The changes from baseline following LYN101 SC administration.
Peak serum concentration (Cmax) | UP to Day 91 in part A. Up to Day 265 in part B
  Cmax of LYN101.
Area under the plasma concentration-time curve from time 0 until the last measurable concentration (AUCtau) of LYN101 | Up to Day 91 in part A. Up to Day 265 in part B.
  AUCtau of LYN101.
Time to cmax (Tmax) of LYN101 | Up to Day 91 in part A. Up to Day 265 in part B.
  Tmax of LYN101
Observed plasma concentration at the end of a dosing interval (Ctrough) of LYN101 | Up to Day 265 in part B.
  Ctrough of LYN101
Terminal Phase Elimination Half-Life (t1/2) of LYN101 | Up to Day 91 in part A. Up to Day 265 in part B.
  T1/2 of LYN101.
Clearance (CL) for LYN101 SC | Up to Day 91 in part A. Up to Day 265 in part B.
  CL for LYN101 SC.
Immunogenicity of LYN101 assessed by anti-drug antibodies (ADAs) | Up to Day 91 in part A. Up to Day 265 in part B.
  Incidence and concentrations of ADAs. Neutralizing ADAs (NAb) may be evaluated.

OTHER OUTCOMES:
Bone mineral density | Up to Day 91 in part A. Up to Day 265 in part B
  The change from baseline after LYN101 or placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Study Director — The First Affiliated Hospital of Bengbu Medical University; Huan Zhou, Dr, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Lin Zhen Zhang, Dr, Principal Investigator — Shanghai 6th People's Hospital
Locations (2):
- China (2):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Shanghai Sixth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No